CLINICAL TRIAL: NCT04380597
Title: Observational and Prospective Study in Patients With Nail Psoriasis Treated With Calcipotriene and Betamethasone Dipropionate Aerosol Foam to Evaluate the Change in the Severity of Psoriasis and in the Quality of Life
Brief Title: Observational Study in Patients With Nail Psoriasis Treated With Enstilar® to Assess the Severity Change and the Quality of Life
Acronym: ENUPS
Status: Completed | Type: Observational
Sponsor: Angeles Florez (Other)
Responsible Party: Sponsor-Investigator, Angeles Florez, Head of Dermatology, Complejo Hospitalario Universitario de Pontevedra
Organization: Complejo Hospitalario Universitario de Pontevedra (Other)
Other Study IDs: ENUPS
Record Dates: First submitted 2019-03-07; First posted 2020-05-08 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2020-05

CONDITIONS: Nail Psoriasis
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Patients with nail psoriasis: Patients with nail psoriasis who are prescribed, according to clinical practice, a topical treatment with calcipotriene and betamethasone dipropionate aerosol foam.
  Interventions: Drug: Calcipotriene and betamethasone dipropionate aerosol foam

INTERVENTIONS:
Drug: Calcipotriene and betamethasone dipropionate aerosol foam — Prescribed according to clinical practice and following Product Data Sheet instructions

SUMMARY:
Observational, prospective and multicentre study to evaluate the effectiveness of calcipotriene and betamethasone dipropionate aerosol foam (Cal / BD), prescribed according to clinical practice and following the Product Data Sheet instructions, in the topical treatment of nail psoriasis according to the change in the score of the Nail Psoriasis Severity Index (NAPSI) at 12 weeks of treatment with respect to the initial score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with nail psoriasis who start, according to clinical practice, topical treatment with calcipotriene and betamethasone dipropionate aerosol foam
* Patients who authorize their participation in the study by signing written informed consent.

Exclusion Criteria:

* Patients receiving treatment with systemic drugs or their prescription is scheduled for the next 3 months. However, may be included patients who receive the same systemic treatment regimen from at least 6 months before their inclusion in the study and up to 14 weeks later.
* Patients with any situation or state that in the opinion of the investigator discourages their participation in the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of nail psoriasis for whom are prescribed, according to clinical practice, a topical treatment. Will be included the first 60 patients that consecutively attend the participating centers and meet all the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Nail Psoriasis Severity Index (NAPSI) | Baseline
  Numeric, reproducible, objective, simple tool for evaluation of nail psoriasis
Nail Psoriasis Severity Index (NAPSI) | Week 12 of treatment
  Numeric, reproducible, objective, simple tool for evaluation of nail psoriasis
Nail Psoriasis Severity Index (NAPSI) | Week 24 of treatment
  Numeric, reproducible, objective, simple tool for evaluation of nail psoriasis

SECONDARY OUTCOMES:
Nail Assessment in Psoriasis and Psoriatic Arthritis (NAPPA) | Baseline, Week 12 of treatment and Week 24 of treatment
  Modular instrument for the assessment of clinical and patient-reported outcomes in nails.

OTHER OUTCOMES:
Hands Photographs | Baseline, Week 12 of treatment and Week 24 of treatment
  High-quality photographs on patient´s both hands to document the psoriasis status

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Pontevedra, Pontevedra, Spain